CLINICAL TRIAL: NCT03667248
Title: Sizing of the PERCEVAL® Sutureless Aortic Valve Prosthesis Using the CT: a Feasibility Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018- 00495; ch18Reuthebuch
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Aortic Valve Stenosis
Keywords: PERCEVAL® sutureless aortic valve prosthesis; aortic valve stenosis; aortic valve replacement; preoperative CT scan of the heart
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sorin Perceval ® Sutureless Valve (Sorin Group Italia Srl, 13040 Saluggia, Italy), available in different sizes (S 19-21mm, M 21-23mm, L 23-25mm, XL 25-27mm) — Sizing of the valve by preoperative CT scan of the heart and comparison of this measurement with the standard procedure (Sizing intraoperatively using the measuring devices provided by the product manufacturer)

SUMMARY:
This study is to analyse if the size of the valve can be determined with a preoperative CT scan of the heart in order to prepare the valve preoperatively to save time.

DETAILED DESCRIPTION:
Patients with severe aortic stenosis undergo aortic valve replacement (AVR). One approach to reduce trauma and operation time is the implantation of a sutureless valve to reduce aortic cross-clamp time due to the missing necessity of suturing the valve. Until now, sizing of the valve was determined intraoperatively using the measuring devices provided by the product manufacturer. Due to the implantation mechanism, the valve has to be collapsed after determination of the size. This is consuming time and can seriously delay the procedure.

This study is to analyse if the size of the valve can be determined with a preoperative CT scan of the heart in order to prepare the valve preoperatively to save time.

ELIGIBILITY:
Inclusion Criteria:

* Implantation of a Sorin Perceval ® sutureless valve
* availability of preoperative CT scan

Exclusion Criteria:

* denial of consent
* missing preoperative CT scan
* bad quality of preoperative CT scan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with implantation of a Sorin Perceval ® sutureless valve at University Hospital Basel/ Switzerland
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
accuracy of aortic valve sizing by preoperative CT scan of the heart | during surgery procedure
  accuracy of aortic valve sizing by preoperative CT scan of the heart in comparison with the standard procedure (Sizing intraoperatively using the measuring devices provided by the product manufacturer)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, PD Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Switzerland